CLINICAL TRIAL: NCT06287060
Title: BLEACHING EFFECT OF STRAWBERRY EXTRACT VERSUS HYDROGEN PEROXIDE IN PATIENTS WITH EXRINSIC STAINING A RANDOMIZED CLINICAL TRIAL
Brief Title: Bleaching Effect of Strawberry Extract Versus Hydrogen Peroxide in Patients With Extrinsic Staining
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Randa Khaled Mostafa, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Strawberry extract
Record Dates: First submitted 2024-02-23; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Bleaching Effect and Postoperative Sensitivity of Strawberry Extract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with extrinsic staining will be treated with strawberry extract. (Experimental)
  Interventions: Other: strawberry extract.
- patients with extrinsic staining will be treated with Hydrogen peroxide bleaching agent. (Active Comparator)
  Interventions: Other: strawberry extract.

INTERVENTIONS:
Other: strawberry extract. — strawberry has a whitening effect due to its content of ellagic and maleic acids. the presence of acidic components namely ascorbic acid may increase the surface energy by removing the surface debris, thereby allowing the citric and maleic acids to penetrate into tooth surface to remove the surface stains.

SUMMARY:
with limited evidence based information in literature about using Strawberry extract for teeth bleaching in patients with extrinsic staining , it is beneficial to evaluate this new material using a randomized controlled clinical trial to test the null hypothesis that this extract will have the same effect as Hydrogen peroxide regarding the bleaching effect and hypersensitivity.

DETAILED DESCRIPTION:
The whitening effect of strawberry is due to the presence of malic acid, which acts as a natural astringent to remove surface discoloration. The ellagic acid content in strawberry is ranging from 0.43 to 4.64 mg/g dry weight. The more amount of ellagic acid will produce more potential OH clusters as a powerful oxidizer thus make the more effective bleaching process. Ellagic acid releases the OH and H radicals which will react with the tooth enamel organic molecules and disrupt the electron conjugation, as well as changing the energy absorption in the tooth enamel organic molecules to form smaller organic molecules with a lighter color. Ellagic acid has an OH cluster, not COOH cluster like any other acids. The electronegativity of the OH group will be easier to break and react with the organic molecules of tooth enamel.

ELIGIBILITY:
Inclusion Criteria:

Participant inclusion criteria:

1. At least 18 years old.
2. Good general and oral health.
3. six present maxillary anterior teeth.

Tooth inclusion criteria:

1. yellowing of teeth due to age.
2. stains due to coffee or tea.
3. light tetracycline stain.

   * Exclusion Criteria:

participant exclusion criteria:

1. patients undergoing radiotherapy or chemotherapy.
2. Pregnant females or breast feeders.
3. Bruxism and patients who reported tooth sensitivity.

Tooth exclusion criteria:

1. Hypoplastic enamel.
2. carious lesion.
3. sensitive recession area or sensitive tooth.
4. Amalgam staining.
5. Non vital tooth.
6. Discolration due to pulp trauma or necrosis.
7. presence of non carious cervical lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Bleaching effect of strawberry extract versus Hydrogen peroxide. | immediately , one week and one month after application.
  objective assessment for the bleaching effect by spectrophotometer.

SECONDARY OUTCOMES:
post operative sensitivity. | immediately after bleaching agent removal , 24 hours after application.
  Tooth sensitivity is scored according to the VRS verbal Rating scale, where 0=none, 1=mild, 2=moderate, 3=considerable, and 4=severe